CLINICAL TRIAL: NCT04437641
Title: Impact of Pediatrician Intervention on the Smoking Habits of Parents of Children With Cystic Fibrosis, Type 1 Diabetes or Children Hospitalized for a First Episode of Bronchiolitis.
Brief Title: Impact of Pediatrician Intervention on the Smoking Habits of Parents of Sick Children
Acronym: MUCODIABTAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/19/0359
Record Dates: First submitted 2020-03-26; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Tobacco Consumption; Bronchiolitis
Keywords: Tobacco Consumption
MeSH Terms: conditions — Tobacco Use; Bronchiolitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: A questionnaire on smoking habits was given to all parents of children being followed in consultation for cystic fibrosis or type 1 diabetes, or whose child was hospitalized for the first time for bronchiolitis.
  Interventions: Other: Tobacco questionnaire

INTERVENTIONS:
Other: Tobacco questionnaire — A questionnaire on smoking habits was given to all parents of children being followed in consultation for cystic fibrosis or type 1 diabetes, or whose child was hospitalized for the first time for bronchiolitis.
  Provision of minimal advice (oral and a leaflet from the anti-smoking centre) to parents who smoke by the paediatrician following the child.
  For parents who smoke, evaluation at 3 months of the impact of this minimal advice by another questionnaire during the usual follow-up of the patient at 3 months or by telephone contact.

SUMMARY:
Reducing tobacco consumption is a major public health objective, with the prevalence of active smoking estimated in 2017 at 26.9% of the French population aged 18 to 25. The negative impact of passive smoking on children's health and development has been demonstrated by numerous studies, especially with regard to respiratory pathologies. Parental smoking is also a risk factor for active smoking in adolescence and adulthood (with an odds ratio of 1.72 if at least one of the two parents is a smoker). It has been shown that intervention with parents can reduce the number of children exposed to passive parental smoking by about 5%.

DETAILED DESCRIPTION:
Reducing tobacco consumption is a major public health objective, with the prevalence of active smoking estimated in 2017 at 26.9% of the French population aged 18 to 25. The negative impact of passive smoking on children's health and development has been demonstrated by numerous studies, especially with regard to respiratory pathologies. Parental smoking is also a risk factor for active smoking in adolescence and adulthood (with an odds ratio of 1.72 if at least one of the two parents is a smoker). It has been shown that intervention with parents can reduce the number of children exposed to passive parental smoking by about 5%. The paediatrician's role is therefore to try to make parents aware of the consequences of tobacco consumption on their children's health and to encourage them to stop smoking. Minimal advice (simple, clear, written and oral information on the actors and means of helping to stop smoking) is the first step in triggering an attempt to stop smoking. The paediatrician seems to be a particularly influential actor since he intervenes at a time when parents are trying to improve their child's health. The minimum advice would have an effectiveness of 2-5% on smoking cessation in general. There is no data on the impact of this minimum advice when given by paediatricians. There are also no data on the current prevalence of smoking in France among parents of children with various chronic diseases, such as cystic fibrosis or diabetes. It is also necessary to describe the smoking habits of parents, as children's exposure and its impact on their health depends in particular on where their parents smoke.

ELIGIBILITY:
Inclusion Criteria:

* Parents of legal age, of children being followed for cystic fibrosis or type 1 diabetes or being hospitalized for the first time for bronchiolitis.
* Having given their non-opposition to participate in the research
* Covered by a social security scheme

Exclusion Criteria:

* Refusal to participate
* Parent already in the process of quitting smoking
* Adult person under guardianship/curators or safeguard of justice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of parents accompanying paediatric patients followed in consultation or seen in hospital in the departments of pneumology and paediatric diabetology at Toulouse University Hospital.
  The doctor proposes to the parent to participate in this research and informs him/her:
  * of the objective,
  * of the computerised processing of the data concerning him/her that will be collected in the course of this research and also specifies his/her rights of access, opposition and rectification to this data.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Smoking prevalence | 18 months
  establish the effect of minimal advice (oral + orientation leaflet) given by the paediatrician following children with cystic fibrosis, diabetes or hospitalized for a first episode of bronchiolitis on the parents' smoking habits.

SECONDARY OUTCOMES:
Parental smoking evolution | 18 months
  Evolution of parental smoking habits 3 months after this advice by :
  Smoking statue number of cigarets/day

CONTACTS AND LOCATIONS:
Overall Officials: Marie MITTAINE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- MITTAINE, Toulouse, France